CLINICAL TRIAL: NCT02569632
Title: Immunogenicity of a U.S.-Licensed Meningococcal Serogroup B Vaccine (Trumenba) in Adults at Increased Risk of Meningococcal Disease Because of Occupational Exposure
Brief Title: Investigating the Immunogenicity of a U.S.-Licensed Meningococcal Serogroup B Vaccine (Trumenba)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UCSF Benioff Children's Hospital Oakland (Other)
Collaborators: University of Massachusetts, Worcester (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ChildrensHRCOakland
Record Dates: First submitted 2015-09-30; First posted 2015-10-07 (Estimated); Results first posted 2021-02-02 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-02

CONDITIONS: Meningococcal Infections
Keywords: Meningococcal Vaccines; Neisseria Meningitidis; Factor H-binding Protein
MeSH Terms: conditions — Meningococcal Infections | interventions — MenB-FHbp vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open Label: MenB-FHbp (Experimental): Trumenba Meningococcal Group B Vaccine (Wyeth/Pfizer Pharmaceuticals)
  Interventions: Biological: Trumenba Vaccine (Wyeth/Pfizer Pharmaceuticals)

INTERVENTIONS:
Biological: Trumenba Vaccine (Wyeth/Pfizer Pharmaceuticals) — All subjects will receive three doses of a Trumenba, a U.S.-licensed meningococcal vaccine. Each 0.5 mL dose contains 60 micrograms of each FHbp variant (total of 120 micrograms of protein), 0.018 mg of PS80 and 0.25 mg of Al³+ as AlPO4 in 10 mM histidine buffered saline at pH 6.0. Trumenba is administered as a three dose series (0.5 mL each) according to a 0-, 2-, and 6-month schedule.
  Other Names: MenB-FHbp

SUMMARY:
This study will investigate the breadth of protection against meningococcal disease in humans immunized with a newly FDA approved meningococcal B vaccine, trade name "Trumenba®" manufactured by Pfizer Vaccines. As a secondary goal the investigators will investigate underlying mechanisms by which human anti-FHbp antibodies elicit complement-mediated bactericidal activity.

DETAILED DESCRIPTION:
Neisseria meningitidis causes meningitis and severe infections of the blood stream. The incidence of serogroup B meningococcal disease however is too low to conduct a randomized, controlled trial to determine the actual efficacy of the new serogroup B vaccines. Instead vaccine efficacy was inferred from serum bactericidal antibody responses using four test strains. However, because of strain variability of FHbp amino acid sequence (there are more than 800 sequence variants described) and strain variability of FHbp expression, bactericidal data on only four strains are unlikely to be sufficient to predict the actual strain coverage by the vaccine. There also are gaps in knowledge about the underlying mechanisms by which human antibodies to FHbp elicit complement mediated bactericidal activity. For example, binding of FH to FHbp is specific for human FH. Therefore in vaccinated humans the vaccine antigen is expected to form a complex with FH right after immunization. The investigators' hypothesis is that binding of human FH to the vaccine antigen skews the antibody repertoire to FHbp epitopes located outside of the FH combining site. The resulting antibodies would be expected not to inhibit binding of FH to the bacteria. This hypothesis will be investigated in Trumenba-immunized humans as part of studies in Aim 1 (and in future studies of recombinant human anti-FHbp Fabs that will be enabled by obtaining DNA from individual B cells, described in Aim 2).

ELIGIBILITY:
Inclusion Criteria:

* Adults in the following risk groups: physicians, nurses, respiratory therapists, microbiology laboratory personnel working at UCSF Benioff Children's Hospital Oakland or the University of Massachusetts Medical School as well as medical students attending accredited U.S. medical schools
* Able to comprehend and follow all required study procedures
* In good health as determined by a brief medical history
* For females of child bearing age a negative urine pregnancy test will be required

Exclusion Criteria:

* Are not in the risk groups summarized above
* Have not given or are unable to give written informed consent to participate in the study
* Females of child bearing potential who are pregnant, or planning on becoming pregnant during the study period.
* Persons with a past history of having Guillain-Barré Syndrome (GBS), or a family history of GBS in a parent or sibling.
* Persons with presence or suspected presence of serious chronic disease including but not limited to: chronic cardiac disease, autoimmune disease, diabetes, hepatitis B/C, HIV, progressive neurological disease or seizure, leukemia, lymphomas, or neoplasm.
* Have participated in any other investigational drug or received any other vaccine within the last 30 days.
* Received a dose of a meningococcal serogroups A, C, Y, W conjugate vaccine within the previous 30 days or wish to receive a dose of this vaccine during the six month study period.
* Have a history of anaphylactic shock, asthma, urticaria or other allergic reaction after previous dose of Trumenba
* Have experienced fever (oral temperature above 38.0°C) within the past 3 days or are suffering from a present acute infectious disease
* Are planning to leave the area of the study site before the end of the study period
* Have obesity (BMI higher than 33); or 11.
* With any condition which, in the opinion of the investigator, might interfere with the evaluation of the study objectives.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dan Granoff, MD, Principal Investigator — Children's Hospital Oakland Research Institute, Center for Immunobiology and Vaccine Development
Locations (2):
- United States (2):
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - University of Massachusetts Medical School, Worcester, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lujan E, Partridge E, Giuntini S, Ram S, Granoff DM. Breadth and Duration of Meningococcal Serum Bactericidal Activity in Health Care Workers and Microbiologists Immunized with the MenB-FHbp Vaccine. Clin Vaccine Immunol. 2017 Aug 4;24(8):e00121-17. doi: 10.1128/CVI.00121-17. Print 2017 Aug. PMID 28566335

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Open Label: MenB-FHbp
Started | 18
Completed | 17
Not Completed | 1

BASELINE CHARACTERISTICS:
Population: The data from one subject enrolled in the study were excluded due to a diagnosis of cancer after dose 2.
Arm/Group | Open Label: MenB-FHbp
Number analyzed (Participants) | 18
Age, Continuous [Median (Full Range); unit: years] | 40 [17 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Breadth of Protective Activity of Serum Anti-FHbp Antibody Responses of Adults Immunized With Trumenba Vaccine as Assessed by Serum Bactericidal Titers
Description: Determine the percentage of subjects achieving serum bactericidal titers of 1:4 or greater in serum obtained 1 month after doses 2 and 3 as measured against a panel of 15 genetically diverse meningococcal strains.
Time Frame: 18 months
Measure: Number; unit: percentage of participants
Arm/Group | Open Label: MenB-FHbp
Number analyzed (Participants) | 17
percentage of participants | 93

2. Secondary Outcome: Antibody Repertoire to FHbp
Description: Determine the percentage of recombinant anti-FHbp Fabs isolated from B cells of each subject that react with 3 FHbp amino acid sequence variants representative of FHbp variant groups 1, 2 and 3
Time Frame: 1 year
Population: This was an exploratory objective requiring new technology. It was done on 0/17 subjects because of technical limitation.
Arm/Group | Open Label: MenB-FHbp
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Open Label: MenB-FHbp
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 1/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label: MenB-FHbp (N=18)
rash (Skin and subcutaneous tissue disorders) | 1 (2) — One subject developed a severe local reactions after doses 1 and 2.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-14): https://cdn.clinicaltrials.gov/large-docs/32/NCT02569632/Prot_SAP_000.pdf